CLINICAL TRIAL: NCT06614491
Title: A Single-Time-Point, Observational Study to Evaluate Interrater Reliability of SACS 2.0 for the Assessment of Peristomal Skin Health in Ostomates
Brief Title: SCOPE - Single-Point Classification Observational Peristomal Evaluation
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OC-24-448
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ileostomy; Colostomy; Urostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ileostomy: Subjects with ileostomy
- Colostomy: Subjects with colostomy
- Urostomy: Subjects with urostomy

SUMMARY:
Study to create an ostomy dataset and collect stoma photos to enable evaluation of images digitally versus an in-person ostomy skin assessment.

DETAILED DESCRIPTION:
The purpose of this study is to create an ostomy dataset and collect stoma photos to enable SACS 2.0 evaluation of images digitally versus an in-person ostomy skin assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ileostomy, colostomy or urostomy
* Age ≥ 18 years of age
* Able and willing to provide informed consent

Exclusion Criteria:

* Enterocutaneous fistulae
* Patients with two or more ostomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 600 Subjects, or 200 Subjects with ileostomy, colostomy, or urostomy peristomal skin categories
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Reliability of SACS assessment | Baseline
  The equivalence of weighted Kappa concordance between SACS assessment via in-person skin assessment by an ostomy care nurse and SACS assessment via examining the skin via photo by a study nurse coordinator

SECONDARY OUTCOMES:
Ostomy dataset | Baseline
  Frequency of peristomal skin health classification scores in 600 consecutive ostomates

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Guerrero, MD, Principal Investigator — Principal Investigator Colombia; Maria Angela Boccara de Paula, PhD, Principal Investigator — Principal Investigator Brazil
Locations (4):
- ConvaCare clinic, São Paulo, Brazil
- Colombia (3):
  - ConvaCare clinic, Bogotá
  - Convacare clinic, Cali
  - ConvaCare clinic, Medellín